CLINICAL TRIAL: NCT00607555
Title: Observational Study on the Effects of Enteral Feeding and Feeding Methods on Respiratory Pattern as Assessed by Diaphragm Electrical Activity (EAdi) in Very Low Birth Weight Preterm Infants
Brief Title: A Study on the Effects of Feeding and Feeding Methods on Breathing Pattern in Very Low Birth Weight Preterm Infants
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Eugene Ng, MD, FRCPC, Sunnybrook Health Sciences Centre
Other Study IDs: 268-2007
Record Dates: First submitted 2008-02-04; First posted 2008-02-05 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2008-09

CONDITIONS: Infant, Premature; Apnea
Keywords: Infant, premature; Infant, very low birth weight; Apnea; Feeding methods; Diaphragm
MeSH Terms: conditions — Premature Birth; Apnea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Premature infants over 23 weeks of gestation and less than 1.25 kilograms at birth, who are tolerating feedings, and are clinically stable
  Interventions: Device: Insertion of specialized feeding tube for monitoring of EAdi

INTERVENTIONS:
Device: Insertion of specialized feeding tube for monitoring of EAdi — The specialized feeding tube will be inserted into the esophagus and positioned at the level of the crural diaphragm. EAdi will be measured with miniaturized coated stainless steel electrodes mounted on the feeding tube. The tube is connected to a monitor where EAdi will be recorded continuously throughout the entire study period

SUMMARY:
In this study, we want to see how feeding affects breathing in small premature babies. Using a special feeding tube in the stomach, we can measure how the diaphragm (a large breathing muscle) might be affected by feeding. We also want to see if slowing down the feeding may lessen this effect.

DETAILED DESCRIPTION:
Premature babies may have pauses in breathing known as apnea, which may require invasive treatment. The exact cause of apnea is unknown, and may be related to a combination of brain, gut, and lung immaturity.

Research in premature babies suggests that feeding may affect lung functions, but such effects may be lessened if feeds are given at a slower rate. Further research showed that the diaphragm, an important breathing muscle, may be fatigued by a full stomach. We speculate that, in premature babies, feeding might tire the diaphragm, thus impairing lung function and possibly causing apnea.

We plan to study 10 stable premature babies less than 23 weeks and 1.25 kilograms at birth. By inserting a special feeding tube with sensors into the stomach, we can measure the electrical activity of the diaphragm (EAdi). By analysing EAdi before and after feeding, we want to directly measure how feeding might affect lung functions. We also want to compare feeding at the usual rate (5-15 minutes) versus a slower rate (90 minutes) to see how their effects on lung functions might differ.

This important study will help us determine the most appropriate treatment for premature babies with apnea related to feeding.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants >23 weeks gestation
* Birth weight <1250 grams
* Not requiring full mechanical ventilation
* Tolerating full regular bolus feeding for at least 48 hours

Exclusion Criteria:

* Congenital and acquired problem of the gastrointestinal tract
* Phrenic nerve injury and/or diaphragm paralysis
* Esophageal perforation/tracheoesophageal fistula
* Congenital/acquired neurological deficit and/or seizures
* Hemodynamic instability
* Congenital heart disease (including symptomatic patent ductus arteriosus)
* Undergoing treatment for sepsis or pneumonia
* Use of muscle relaxants, narcotic analgesics, or gastric motility agents

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants admitted to the Neonatal Intensive Care Unit of Sunnybrook Health Sciences Centre
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in amount of tonic electrical activity of the diaphragm (EAdi) from baseline during and after an intermittent bolus feed | Day of study

SECONDARY OUTCOMES:
Change in amount of phasic EAdi before and after an intermittent bolus feed | Day of study
Change in the number of apnea episodes on the EAdi waveform before and after an intermittent bolus feed | Day of study
Changes in tonic and phasic EAdi, and apnea between intermittent bolus and intermittent slow-bolus feed | Day of study
Diaphragmatic fatigue | Day of study
Episodes of clinically significant apnea between intermittent bolus and intermittent slow bolus feed | Day of study
Episodes of regurgitation or vomiting between intermittent bolus and intermittent slow bolus feed | Day of study

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Ng, MD, FRCPC, Study Chair — Sunnybrook Health Sciences Centre; Patti Schurr, RN, MSc, Principal Investigator — Sunnybrook Health Sciences Centre; Maureen Reilly, RRT, Principal Investigator — Sunnybrook Health Sciences Centre; Jennifer Beck, PhD, Study Director — Sunnybrook Health Sciences Centre; Michael Dunn, MD, FRCPC, Study Director — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada